CLINICAL TRIAL: NCT06636955
Title: Viral Epidemiology of Bronchiolitis After NIrsevimab Implementation and Respiratory Evolution in Infants
Acronym: EBINIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0184/HP; 2024-A01498-39 (Registry Identifier: ID RCB)
Record Dates: First submitted 2024-09-19; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Bronchiolitis
Keywords: Nirsevimab; passive immunization; pediatric emergencies; viral epidemiology; acute bronchilitis
MeSH Terms: interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * nasopharyngeal swabs
  * nasal enema
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- passive immunization: Patients having received a passive immunization
  Interventions: Other: biobank; Other: follow up
- no passive immunization: Patients not having received a passive immunization
  Interventions: Other: biobank; Other: follow up

INTERVENTIONS:
Other: biobank — * nasopharyngeal swab collection
  * nasopharyngeal nasal washes collection, during hospitalization, if any
Other: follow up — - one year follow up: after 1 month, 3 months, 6 months et 12 months

SUMMARY:
Acute bronchiolitis in infants, mainly caused by the Respiratory Syncytial Virus (RSV), is a public health issue, in terms of morbidity and hospital costs.

Nirsevimab, a long-acting antibody against RSV available for all infants under 12 months, could profoundly modify the epidemiology of the next epidemic seasons, with the increase of the frequency of the other respiratory viruses (endemic Coronaviruses, Metapneumovirus, etc) Monitoring viral ecology is important, as the impact of respiratory infections on morbidity in the short, medium and long term, but also in economic terms.

Infants under the age 12 months with a first episode of bronchiolitis and consulting the emergency pediatric department will be included. A nasopharyngeal swab will be performed as routine care, and clinical data will be collected.

Multiplex Polymerase Chain Reaction will be performed to identify respiratory virus(es) responsible for the bronchiolitis. In hospitalized infants with RSV or rhinovirus positive Polymerase Chain Reaction (PCR), daily nasal washes will be collected to perform viral loads with specific quantitative PCR (nasal washes biobank), associated with daily clinical data. A 12-month follow-up is planned for every infant included, consisting with 4 phone calls, to identify factors associated with the onset of preschool wheezing.

The main objective is to describe the viral epidemiology associated with acute bronchiolitis leading to a pediatric emergency department visit the implementation of Nirsevimab.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 12 months or less
* Admitted to the pediatric emergencies services during one of the three epidemic years: 2024-2025, 2025-2026 and 2026-2027
* With clinical diagnosis of first episode of acute bronchiolitis by the emergency pediatrician
* With nasopharyngeal swab for virological diagnosis

Exclusion Criteria:

* Refusal of one or more of the infants parents to participate in the study
* Infants parents refused to be called back for follow-up
* No nasopharyngeal swab taken

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant with acute bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-10-07 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the prevalence of viral populations identified by respiratory multiplex PCR ( nasopharyngeal swab) in the group with Nirsevimab and in the group without Nirsevimab | 3 years
  Multiplex Polymerase Chain Reaction (nasopharyngeal swab) in the 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No